CLINICAL TRIAL: NCT01626157
Title: A Novel Assay to Quantify Treatment Response in CF
Brief Title: A Novel Assay to Quantify Treatment Response in Cystic Fibrosis (CF)
Status: Completed | Type: Observational
Sponsor: Milene Saavedra (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor-Investigator, Milene Saavedra, Assistant Professor, National Jewish Health
Organization: National Jewish Health (Other)
Other Study IDs: SAAVED11A0
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inflammation is present in the Cystic fibrosis (CF) airway from the time of infancy, and worsens with the onset of chronic infection. Therapies with proven benefit are associated with decreased airway inflammation. Thus, sensitive and reproducible biomarkers of airway inflammation have long been sought as a necessary component to improved clinical care and to facilitate therapeutic trials for CF. FEV1, the standard outcome measure in CF, is recognized as an insensitive outcome measure. the investigators have identified a panel of 10 genes which sensitively predict resolution of pulmonary inflammation, in response to therapy of an acute pulmonary exacerbation. With the goal of yielding a technically simple but unique CF biomarker assay, the investigators have tested whether proteins signified by these genes show large changes in expression following treatment of acute pulmonary exacerbations. Protein quantifications are among the most common measurements performed in clinical laboratories around the world. Based on preliminary findings that changes in white blood cell proteins mirror changes seen in the genes, the investigators propose to identify top candidate proteins, from the investigators gene panel, which change in response to exacerbation therapy. Once identified, these proteins will be quantified directly with a new blood test which is inexpensive and simple to perform. The investigators propose to validate this blood test in a single site trial. If successful, this proposal will yield a biomarker assay that will be available to validate in a multi-site trial and provide unique insights into mechanisms that regulate white blood cell activation and recruitment in CF lung disease.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of CF.
2. Age 18 years old or greater.
3. Presentation at the start of treatment for a pulmonary exacerbation of CF.
4. Ability to perform reproducible Pulmonary Function Tests and produce sputum.
5. Willingness to comply with study procedure and willingness to provide written consent.

Exclusion Criteria:

1. Presence of a condition or abnormality that, in the opinion of the Principal Investigator (PI), would compromise the safety of the patient or the quality of the data.
2. Use of systemic steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult CF patients > 18 years of age undergoing treatment for acute pulmonary exacerbation
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2011-05; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in leukocyte associated protein expression by flow cytometry and by leukocyte specific ELISA in response to acute exacerbation therapy | 10-21 days

SECONDARY OUTCOMES:
Change in FEV1 in response to acute exacerbation therapy | 10-21 days
Change in sputum IL-8 and neutrophil elastase in response to acute exacerbation therapy | 10-21 days
Change in bacterial density in response to exacerbation therapy | 10-21 days
Change in CRP in response to acute exacerbation therapy | 10-21 days
Time to next exacerbation | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Milene Saavedra, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No